CLINICAL TRIAL: NCT06328452
Title: Risk Factors and Impact of Metabolic Dysfunction -Associated Steatotic Liver Disease in Patients With Inflammatory Bowel Disease
Brief Title: Risk Factors and Impact MASLD in Patients With IBD
Acronym: MASLD
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Zeinab Nasr El Din Ahmed, Assistant lecturer, Assiut University
Other Study IDs: MASLD
Record Dates: First submitted 2024-03-16; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Metabolic Dysfunction-associated Steatotic Liver Disease
Keywords: MASLD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: FibroScan — All the study population will be submitted to Fibroscan examination with CAP (Echosens FibroScan® Compact 530). To evaluate steatosis and fibrosis, participants will be asked to fast for at least 3 hours before the test. To capture a controlled attenuation parameter (CAP) score and liver stiffness measurement (LSM), 10 valid scans per subject will be needed.

SUMMARY:
Inflammatory bowel disease (IBD) is a chronic disease characterized by remitting and relapsing inflammation of the gastrointestinal tract. Crohn's disease (CD) and ulcerative colitis (UC) are the two main types of IBD and their incidence and prevalence are increasing.

In about 5-50% of patients with IBD, there are several extraintestinal manifestations as primary sclerosing cholangitis, autoimmune/granulomatous hepatitis, and non-alcoholic fatty liver disease (NAFLD).

Metabolic dysfunction-associated steatotic liver disease "MASLD"(formerly NAFLD) is a spectrum of hepatic diseases associated with metabolic and cardiovascular disorders, such as obesity, insulin resistance (IR), hypertension, dyslipidemia, impaired glucose tolerance and type 2 diabetes mellitus.

The risk factors of developing liver steatosis in patients with IBD remain undetermined. Some studies have supported traditional risk factors, such as type 2 Diabetes mellitus (T2DM), weight gain, or obesity, to contribute to MAFLD development in patients with IBD. Other studies have highlighted the involvement of disease activity, duration, drug-induced liver injury and small bowel surgeries in MAFLD progression.

Limited data are available on the frequency and risk factors of MASLD in Egyptian patients with IBD, and no published Egyptian study has addressed the clinical utility of serum steatosis markers in MASLD prediction in IBD population. Moreover, the impact of MASLD on IBD course is unclear. Therefore, we will conduct our study to shed some light on this issue.

DETAILED DESCRIPTION:
Inflammatory bowel diseases (IBD) are chronic diseases characterized by remitting and relapsing inflammation of the gastrointestinal tract, with negative effects on the patients' social function and quality of life. Crohn's disease (CD) and ulcerative colitis (UC) are the two main types of IBD that present specific characteristics and their incidence and prevalence are globally increasing.

In about 5-50% of patients with IBD, there are several extraintestinal manifestations such as musculoskeletal, ocular, cutaneous, and hepatobiliary. Hepatobiliary manifestations include primary sclerosing cholangitis, autoimmune/granulomatous hepatitis, and in particular, non-alcoholic fatty liver disease (NAFLD).

NAFLD currently the most common chronic liver disease worldwide. Its global prevalence increased over 3 decades from 25.3% to 38%.

NAFLD is a spectrum of hepatic diseases associated with metabolic and cardiovascular disorders, such as obesity, insulin resistance (IR), hypertension, dyslipidemia, impaired glucose tolerance and type 2 diabetes mellitus. It is frequently recognized as the hepatic manifestation of metabolic syndrome.

Therefore, a new broader nomenclature has been introduced that is "Metabolic Dysfunction-associated Fatty Liver Disease" (MAFLD). More recently, a multi society Delphic consensus statement on a new nomenclature of fatty liver disease was published, introducing the term "Metabolic Dysfunction- associated Steatotic Liver Disease (MASLD) to make the term NAFLD retired.

Estimates of liver steatosis prevalence in IBD patients vary widely from 8% to 88%. This could be explained by heterogeneity of the diagnostic methods and the selected study population.

The risk factors of developing liver steatosis in patients with IBD remain undetermined. Some studies have supported traditional risk factors, such as type 2 Diabetes mellitus (T2DM), weight gain, or obesity, to contribute to MAFLD development in patients with IBD. Other studies have highlighted the involvement of disease activity, duration, drug-induced liver injury and small bowel surgeries in MAFLD progression.

Several serum scores (biomarkers) have been developed to predict the presence or absence of hepatic steatosis. These scores have been extensively validated both for the general population and obese population. However, little is known about their usefulness in prediction of steatosis in IBD patients.

IBD and fatty liver disease are both associated with considerable healthcare expenditures, and their increasing prevalence would undoubtedly impose a growing economic burden. Moreover, IBD patients with concurrent fatty liver disease are potentially at a higher risk of liver abnormalities compared with those without, which can affect the clinical management of the patients with IBD.

Soni reported greater mortality, morbidity and health care resources utilization in patients with IBD who were hospitalized with concomitant diagnosis of NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will be older than 18 years with an IBD diagnosis according to clinical, laboratory, endoscopic and histopathological evaluation (according to European Crohn's and Colitis Organization (ECCO)) (Maaser et al., 2019)

Exclusion Criteria:

* IBD patients with any of the following conditions will be excluded:

  1. Patients with a history of alcohol or drug abuse
  2. Patients with HCV or HBV infection
  3. Patients with autoimmune liver disease
  4. Hepatic malignancies (primary or secondary)
  5. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This will be a prospective cohort study, conducted in Al Rajhi University Hospital, Assiut University from April 2024 till October 2025. The study population will be recruited from patients attending the IBD Outpatient Clinic and will be categorized into two groups (IBD with MASLD and IBD without MASLD).
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Assess the prevalence and risk factors of metabolic dysfunction associated steatotic liver disease among patients attending inflammatory bowel disease outpatient clinic | 3 months from 1st April to 30th June 2024
  Assess the prevalence and risk factors of metabolic dysfunction associated steatotic liver disease among patients attending inflammatory bowel disease outpatient clinic
Effect of metabolic dysfunction associated steatotic liver disease on inflammatory bowel disease course | from 1st April 2024 to 30th June 2025
  Effect of metabolic dysfunction associated steatotic liver disease on inflammatory bowel disease course (the rate of clinical relapse that will be defined as any occurence of IBD-related admission, surgery, as well as the first use of corticosteroids, immunomodulators or biological agents (either bio-naive or bio-experienced patients) during follow up.

SECONDARY OUTCOMES:
Performance of serum steatosis markers in prediction of steatosis | from 1st April 2024 to 30th June 2025
  Serum steatosis markers: hepatic steatosis index (8 x (ALT/AST ratio) + BMI ( weight and height will be combined to report BMI in kg/m^2) (+2, if female; +2, if diabetes mellitus) will be calculated.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams LC, Lubbe F, Bressem K, Wagner M, Hamm B, Makowski MR. Non-alcoholic fatty liver disease in underweight patients with inflammatory bowel disease: A case-control study. PLoS One. 2018 Nov 14;13(11):e0206450. doi: 10.1371/journal.pone.0206450. eCollection 2018. PMID 30427909
- [Background] Ali MaEH, Kamal GM, Younis MaA, et al. Diagnostic performance of serum steatosis biomarkers in Prediction of Non Alcoholic Fatty Liver Disease in Adult Asymptomatic Egyptians. SVU-International Journal of Medical Sciences, (2022); 5(2): 51-63.
- [Background] Allen AM, Van Houten HK, Sangaralingham LR, Talwalkar JA, McCoy RG. Healthcare Cost and Utilization in Nonalcoholic Fatty Liver Disease: Real-World Data From a Large U.S. Claims Database. Hepatology. 2018 Dec;68(6):2230-2238. doi: 10.1002/hep.30094. Epub 2018 Sep 20. PMID 29774589
- [Background] Barberio B, Zamani M, Black CJ, Savarino EV, Ford AC. Prevalence of symptoms of anxiety and depression in patients with inflammatory bowel disease: a systematic review and meta-analysis. Lancet Gastroenterol Hepatol. 2021 May;6(5):359-370. doi: 10.1016/S2468-1253(21)00014-5. Epub 2021 Mar 12. PMID 33721557
- [Background] Buzzetti E, Pinzani M, Tsochatzis EA. The multiple-hit pathogenesis of non-alcoholic fatty liver disease (NAFLD). Metabolism. 2016 Aug;65(8):1038-48. doi: 10.1016/j.metabol.2015.12.012. Epub 2016 Jan 4. PMID 26823198
- [Background] Cai W, Cagan A, He Z, Ananthakrishnan AN. A Phenome-Wide Analysis of Healthcare Costs Associated with Inflammatory Bowel Diseases. Dig Dis Sci. 2021 Mar;66(3):760-767. doi: 10.1007/s10620-020-06329-9. Epub 2020 May 20. PMID 32436120
- [Background] Capela TL, Silva VM, Freitas M, Arieira C, Goncalves TC, de Castro FD, Magalhaes J, Cotter J. Identifying inflammatory bowel disease patients at risk of metabolic dysfunction-associated fatty liver disease: usefulness of non-invasive steatosis predictive scores. BMC Gastroenterol. 2023 Dec 13;23(1):437. doi: 10.1186/s12876-023-02988-w. PMID 38093213
- [Background] Eslam M, Newsome PN, Sarin SK, Anstee QM, Targher G, Romero-Gomez M, Zelber-Sagi S, Wai-Sun Wong V, Dufour JF, Schattenberg JM, Kawaguchi T, Arrese M, Valenti L, Shiha G, Tiribelli C, Yki-Jarvinen H, Fan JG, Gronbaek H, Yilmaz Y, Cortez-Pinto H, Oliveira CP, Bedossa P, Adams LA, Zheng MH, Fouad Y, Chan WK, Mendez-Sanchez N, Ahn SH, Castera L, Bugianesi E, Ratziu V, George J. A new definition for metabolic dysfunction-associated fatty liver disease: An international expert consensus statement. J Hepatol. 2020 Jul;73(1):202-209. doi: 10.1016/j.jhep.2020.03.039. Epub 2020 Apr 8. PMID 32278004
- [Background] Haas L, Chevalier R, Major BT, Enders F, Kumar S, Tung J. Biologic Agents Are Associated with Excessive Weight Gain in Children with Inflammatory Bowel Disease. Dig Dis Sci. 2017 Nov;62(11):3110-3116. doi: 10.1007/s10620-017-4745-1. Epub 2017 Sep 11. PMID 28895012
- [Background] Hsiao SW, Chen TC, Su PY, Yang CT, Huang SP, Chen YY, Yen HH. Metabolic Dysfunction-Associated Fatty Liver Disease in Taiwanese Patients with Inflammatory Bowel Disease: A Study in Patients with Clinical Remission. Diagnostics (Basel). 2023 Oct 20;13(20):3268. doi: 10.3390/diagnostics13203268. PMID 37892089
- [Background] Keys A, Fidanza F, Karvonen MJ, Kimura N, Taylor HL. Indices of relative weight and obesity. J Chronic Dis. 1972 Jul 1;25(6):329-43. doi: 10.1016/0021-9681(72)90027-6. No abstract available. PMID 4650929
- [Background] Lapumnuaypol K, Kanjanahattakij N, Pisarcik D, Thongprayoon C, Wijarnpreecha K, Cheungpasitporn W. Effects of inflammatory bowel disease treatment on the risk of nonalcoholic fatty liver disease: a meta-analysis. Eur J Gastroenterol Hepatol. 2018 Aug;30(8):854-860. doi: 10.1097/MEG.0000000000001144. PMID 29697458
- [Background] Maaser C, Sturm A, Vavricka SR, Kucharzik T, Fiorino G, Annese V, Calabrese E, Baumgart DC, Bettenworth D, Borralho Nunes P, Burisch J, Castiglione F, Eliakim R, Ellul P, Gonzalez-Lama Y, Gordon H, Halligan S, Katsanos K, Kopylov U, Kotze PG, Krustins E, Laghi A, Limdi JK, Rieder F, Rimola J, Taylor SA, Tolan D, van Rheenen P, Verstockt B, Stoker J; European Crohn's and Colitis Organisation [ECCO] and the European Society of Gastrointestinal and Abdominal Radiology [ESGAR]. ECCO-ESGAR Guideline for Diagnostic Assessment in IBD Part 1: Initial diagnosis, monitoring of known IBD, detection of complications. J Crohns Colitis. 2019 Feb 1;13(2):144-164. doi: 10.1093/ecco-jcc/jjy113. No abstract available. PMID 30137275
- [Background] Magri S, Paduano D, Chicco F, Cingolani A, Farris C, Delogu G, Tumbarello F, Lai M, Melis A, Casula L, Fantini MC, Usai P. Nonalcoholic fatty liver disease in patients with inflammatory bowel disease: Beyond the natural history. World J Gastroenterol. 2019 Oct 7;25(37):5676-5686. doi: 10.3748/wjg.v25.i37.5676. PMID 31602167
- [Background] Malik TF, Aurelio DM. Extraintestinal Manifestations of Inflammatory Bowel Disease. 2023 Mar 6. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK568797/ PMID 33760556
- [Background] Marotto D, Atzeni F, Ardizzone S, Monteleone G, Giorgi V, Sarzi-Puttini P. Extra-intestinal manifestations of inflammatory bowel diseases. Pharmacol Res. 2020 Nov;161:105206. doi: 10.1016/j.phrs.2020.105206. Epub 2020 Sep 28. PMID 32998068
- [Background] Matsuoka K, Kobayashi T, Ueno F, Matsui T, Hirai F, Inoue N, Kato J, Kobayashi K, Kobayashi K, Koganei K, Kunisaki R, Motoya S, Nagahori M, Nakase H, Omata F, Saruta M, Watanabe T, Tanaka T, Kanai T, Noguchi Y, Takahashi KI, Watanabe K, Hibi T, Suzuki Y, Watanabe M, Sugano K, Shimosegawa T. Evidence-based clinical practice guidelines for inflammatory bowel disease. J Gastroenterol. 2018 Mar;53(3):305-353. doi: 10.1007/s00535-018-1439-1. Epub 2018 Feb 10. PMID 29429045
- [Background] Matthews DR, Hosker JP, Rudenski AS, Naylor BA, Treacher DF, Turner RC. Homeostasis model assessment: insulin resistance and beta-cell function from fasting plasma glucose and insulin concentrations in man. Diabetologia. 1985 Jul;28(7):412-9. doi: 10.1007/BF00280883. PMID 3899825
- [Background] Ng SC, Shi HY, Hamidi N, Underwood FE, Tang W, Benchimol EI, Panaccione R, Ghosh S, Wu JCY, Chan FKL, Sung JJY, Kaplan GG. Worldwide incidence and prevalence of inflammatory bowel disease in the 21st century: a systematic review of population-based studies. Lancet. 2017 Dec 23;390(10114):2769-2778. doi: 10.1016/S0140-6736(17)32448-0. Epub 2017 Oct 16. PMID 29050646
- [Background] Rinella ME, Lazarus JV, Ratziu V, Francque SM, Sanyal AJ, Kanwal F, Romero D, Abdelmalek MF, Anstee QM, Arab JP, Arrese M, Bataller R, Beuers U, Boursier J, Bugianesi E, Byrne CD, Narro GEC, Chowdhury A, Cortez-Pinto H, Cryer DR, Cusi K, El-Kassas M, Klein S, Eskridge W, Fan J, Gawrieh S, Guy CD, Harrison SA, Kim SU, Koot BG, Korenjak M, Kowdley KV, Lacaille F, Loomba R, Mitchell-Thain R, Morgan TR, Powell EE, Roden M, Romero-Gomez M, Silva M, Singh SP, Sookoian SC, Spearman CW, Tiniakos D, Valenti L, Vos MB, Wong VW, Xanthakos S, Yilmaz Y, Younossi Z, Hobbs A, Villota-Rivas M, Newsome PN; NAFLD Nomenclature consensus group. A multisociety Delphi consensus statement on new fatty liver disease nomenclature. Ann Hepatol. 2024 Jan-Feb;29(1):101133. doi: 10.1016/j.aohep.2023.101133. Epub 2023 Jun 24. PMID 37364816
- [Background] Ritaccio G, Stoleru G, Abutaleb A, Cross RK, Shetty K, Sakiani S, Wong U. Nonalcoholic Fatty Liver Disease Is Common in IBD Patients However Progression to Hepatic Fibrosis by Noninvasive Markers Is Rare. Dig Dis Sci. 2021 Sep;66(9):3186-3191. doi: 10.1007/s10620-020-06588-6. Epub 2020 Sep 7. PMID 32894439
- [Background] Rodriguez-Duque JC, Calleja JL, Iruzubieta P, Hernandez-Conde M, Rivas-Rivas C, Vera MI, Garcia MJ, Pascual M, Castro B, Garcia-Blanco A, Garcia-Nieto E, Olmo SC, Cagigal ML, Lopez-Montejo L, Fernandez-Lamas T, Rasines L, Fortea JI, Vaque JP, Frias Y, Rivero M, Arias-Loste MT, Crespo J. Increased risk of MAFLD and Liver Fibrosis in Inflammatory Bowel Disease Independent of Classic Metabolic Risk Factors. Clin Gastroenterol Hepatol. 2023 Feb;21(2):406-414.e7. doi: 10.1016/j.cgh.2022.01.039. Epub 2022 Feb 3. PMID 35124272
- [Background] Schroder T, Schmidt KJ, Olsen V, Moller S, Mackenroth T, Sina C, Lehnert H, Fellermann K, Buning J. Liver steatosis is a risk factor for hepatotoxicity in patients with inflammatory bowel disease under immunosuppressive treatment. Eur J Gastroenterol Hepatol. 2015 Jun;27(6):698-704. doi: 10.1097/MEG.0000000000000350. PMID 25923946
- [Background] Sourianarayanane A, Garg G, Smith TH, Butt MI, McCullough AJ, Shen B. Risk factors of non-alcoholic fatty liver disease in patients with inflammatory bowel disease. J Crohns Colitis. 2013 Sep;7(8):e279-85. doi: 10.1016/j.crohns.2012.10.015. Epub 2012 Nov 15. PMID 23158500
- [Background] Theel W, Boxma-de Klerk BM, Dirksmeier-Harinck F, van Rossum EFC, Kanhai DA, Apers J, van Dalen BM, de Knegt RJ, Holleboom AG, Tushuizen ME, Grobbee DE, Wiebolt J, Castro Cabezas M. Evaluation of nonalcoholic fatty liver disease (NAFLD) in severe obesity using noninvasive tests and imaging techniques. Obes Rev. 2022 Aug;23(8):e13481. doi: 10.1111/obr.13481. Epub 2022 Jun 12. PMID 35692179
- [Background] WHO Expert Consultation. Appropriate body-mass index for Asian populations and its implications for policy and intervention strategies. Lancet. 2004 Jan 10;363(9403):157-63. doi: 10.1016/S0140-6736(03)15268-3. PMID 14726171
- [Background] Yen HH, Su PY, Huang SP, Wu L, Hsu TC, Zeng YH, Chen YY. Evaluation of non-alcoholic fatty liver disease in patients with inflammatory bowel disease using controlled attenuation parameter technology: A Taiwanese retrospective cohort study. PLoS One. 2021 May 27;16(5):e0252286. doi: 10.1371/journal.pone.0252286. eCollection 2021. PMID 34043691
- [Background] Younossi ZM, Golabi P, Paik JM, Henry A, Van Dongen C, Henry L. The global epidemiology of nonalcoholic fatty liver disease (NAFLD) and nonalcoholic steatohepatitis (NASH): a systematic review. Hepatology. 2023 Apr 1;77(4):1335-1347. doi: 10.1097/HEP.0000000000000004. Epub 2023 Jan 3. PMID 36626630
- [Background] Younossi ZM, Koenig AB, Abdelatif D, Fazel Y, Henry L, Wymer M. Global epidemiology of nonalcoholic fatty liver disease-Meta-analytic assessment of prevalence, incidence, and outcomes. Hepatology. 2016 Jul;64(1):73-84. doi: 10.1002/hep.28431. Epub 2016 Feb 22. PMID 26707365
- [Background] Zamani M, Alizadeh-Tabari S, Singh S, Loomba R. Meta-analysis: prevalence of, and risk factors for, non-alcoholic fatty liver disease in patients with inflammatory bowel disease. Aliment Pharmacol Ther. 2022 Apr;55(8):894-907. doi: 10.1111/apt.16879. Epub 2022 Mar 11. PMID 35274325
- [Background] Zou ZY, Shen B, Fan JG. Systematic Review With Meta-analysis: Epidemiology of Nonalcoholic Fatty Liver Disease in Patients With Inflammatory Bowel Disease. Inflamm Bowel Dis. 2019 Oct 18;25(11):1764-1772. doi: 10.1093/ibd/izz043. PMID 30918952